CLINICAL TRIAL: NCT05781724
Title: Cardiac Biomarkers:Comparison Between Analytical Methods
Brief Title: Cardiac Biomarkers and Analytical Methods
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Baroni Silvia, Confirmed researcher - Adjunct Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2216
Record Dates: First submitted 2023-02-21; First posted 2023-03-23 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Diseases; Myocardial Injury
Keywords: Troponin; sST2; NT-ProBNP; Laboratory assay
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — residual serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the western world the prevalence of myocardial infarction is estimated at around 1-2% of the population; increases progressively with age, reaching a percentage of 10% after the 75 years.

It is therefore considered the first cause of hospitalization and mortality in Western countries, as well as expenditure for the health system.

It is therefore very important to have cardiac biomarkers that allow to confirm the diagnostic suspicion of coronary heart disease and/or heart failure, carry out prognostic evaluations and stratify patients as precisely as possible in relation to their actual risk.

Currently as biomarkers of heart failure, natriuretic peptides (BNP and NT-proBNP) are widely used in clinical practice but, considering the complexity of heart failure and its clinical and pathophysiological heterogeneity, it is reasonable to think that a single biomarker is not sufficient . For these reasons, there is increasing interest in the scientific community in the search for new biomarkers useful for early diagnosis, for correct prognostic stratification and for evaluating the response to therapy.

DETAILED DESCRIPTION:
The study aims to evaluate the analytical performance of different kits and molecular markers commercially available (or in pre-industrial development phase) for the assays of the cardiac biomarkers: cTnI , NT-proBNP and sST2.

500 samples (residual serum) from patients hospitalized and/or referred to the DEA Department, for which troponin and/or NT-proBNP tests have been requested routinely or urgently by clinicians, will be included in the study.

The analytical performance of the various kits and the intra- and interassay imprecision will be evaluated. Comparison of methods will be calculated by Passing-Bablok regression and graph by Bland-Altman.

Through the non-parametric Passing-Bablok model the obtained data will be compared with the various analytical methods, reporting them one in function of the other, together with the regression line.

From the regression equation, the proportional systematic error will be evaluated as angular coefficient of the straight line and the constant systematic error as an intercept of the equation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients arriving in the emergency room with chest pain of presumable cardiac origin and uncertain etiological diagnosis
* Routine request for cardiac Troponin and NT-ProBNP

Exclusion Criteria:

* Age <18 years;
* No requirement for cardiac Troponin and NT-ProBNP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 samples, of residual serum, from patients hospitalized and/or referred to the DEA of our Polyclinic, for which troponin and/or NT-proBNP tests have been requested routinely or urgently by clinicians, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate current and new laboratory methods and assays | 24 months
  The analytical performance of the assay will be evaluated according to the Clinical and Laboratory Standards Institute (CLSI) EP15-A3 guidelines with the aim to highlight the differences respect to the methods currently used in laboratory and optimize the diagnostic accuracy and precison of the available tests.
  Comparison between different methods with different analytical sensitivity for the same cardiac biomarker (eg Troponin ultra- Troponin Singulex- Troponin Hs).
Evaluate new cardiac biomarkers | 24 months
  Evaluate new cardiac biomarkers (eg sST2) to implement in the panel of available assays, in response to clinician requests, international guidelines and the emerging potential of new biochemical tests.
  Evaluate the medium-long term (1 year) predictive value of the new biomarker in the heart patients attending at the Emergency Department for non-STEMI Acute Chest Pain.

SECONDARY OUTCOMES:
Create a multiparametric algorithm/score | 36 months
  Integrate the new cardiac biomarkers values in a multiparametric algorithm/score for the differential diagnosis and risk stratification in medium/long-term complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Baroni, Roma, Italy

REFERENCES:
- [Background] Apple FS, Collinson PO; IFCC Task Force on Clinical Applications of Cardiac Biomarkers. Analytical characteristics of high-sensitivity cardiac troponin assays. Clin Chem. 2012 Jan;58(1):54-61. doi: 10.1373/clinchem.2011.165795. Epub 2011 Sep 30. PMID 21965555
- [Background] Bonaca MP, Ruff CT, Kosowsky J, Conrad MJ, Murphy SA, Sabatine MS, Jarolim P, Morrow DA. Evaluation of the diagnostic performance of current and next-generation assays for cardiac troponin I in the BWH-TIMI ED Chest Pain Study. Eur Heart J Acute Cardiovasc Care. 2013 Sep;2(3):195-202. doi: 10.1177/2048872613486249. PMID 24222830
- [Background] Januzzi JL, Mebazaa A, Di Somma S. ST2 and prognosis in acutely decompensated heart failure: the International ST2 Consensus Panel. Am J Cardiol. 2015 Apr 2;115(7 Suppl):26B-31B. doi: 10.1016/j.amjcard.2015.01.037. Epub 2015 Jan 23. PMID 25665762
- [Background] Samaha E, Avila A, Helwani MA, Ben Abdallah A, Jaffe AS, Scott MG, Nagele P. High-Sensitivity Cardiac Troponin After Cardiac Stress Test: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2019 Mar 19;8(6):e008626. doi: 10.1161/JAHA.118.008626. PMID 30871395
- [Background] Neumann JT, Havulinna AS, Zeller T, Appelbaum S, Kunnas T, Nikkari S, Jousilahti P, Blankenberg S, Sydow K, Salomaa V. Comparison of three troponins as predictors of future cardiovascular events--prospective results from the FINRISK and BiomaCaRE studies. PLoS One. 2014 Mar 4;9(3):e90063. doi: 10.1371/journal.pone.0090063. eCollection 2014. PMID 24594734
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Result] Sarlo F, De Luca C, Moretti G, Urbani A, Baroni S. Analytical performance evaluation of the new sST2 turbidimetric assay implemented in laboratory automation systems. Clin Chem Lab Med. 2021 Oct 18;60(2):e54-e56. doi: 10.1515/cclm-2021-0851. Print 2022 Jan 27. No abstract available. PMID 34655512